CLINICAL TRIAL: NCT04738890
Title: Online Mindfulness-based Cognitive Therapy for Parents of Children With Food Allergies: A Pilot Randomised Control Trial.
Brief Title: Online Mindfulness-based Cognitive Therapy for Parents of Children With Food Allergies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EllieCraig2021
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2022-03

CONDITIONS: The Quality of Life of Parents of Children With Food Allergy
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCT-PCCFA plus TAU (Experimental): Mindfulness-based cognitive therapy adapted for parents and carers of children with food allergy (MBCT-PCCFA) offered live online by video-conferencing, plus treatment as usual.
  Interventions: Behavioral: Mindfulness-based cognitive therapy; Other: Treatment as usual
- TAU control (Other): Treatment as usual control group
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy — Mindfulness-based cognitive therapy adapted for parents and carers of children with food allergy (MBCT-PCCFA) offered live online by video-conferencing
  Arms: MBCT-PCCFA plus TAU
Other: Treatment as usual — Continuance as planned of whatever other treatments or interventions the participants were receiving at the time of recruitment.

SUMMARY:
This study aims to conduct an initial evaluation of adapted, live online, mindfulness-based cognitive therapy for parents and carers of children with food allergies (MBCT-PCCFA).

DETAILED DESCRIPTION:
This study is a pilot randomised controlled trial (RCT) comparing adapted, live online, mindfulness-based cognitive therapy for parents and carers of children with food allergies (MBCT-PCCFA) with a treatment as usual control. A battery of self-report measures will be administered online at baseline (week 0), post-intervention (week 15) and at follow-up (week 23).

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregivers who identify as having a child under the age of 18 with a food allergy
* The allergy has been diagnosed by a qualified physician (e.g. GP or allergy specialist)
* Mean score of >=2 on the FAQL-PB, indicating they are at least 'somewhat limited/troubled' by their child's allergy (Cohen et al., 2004).
* Resident in the United Kingdom
* Have access to email, a PC/laptop/tablet with a webcam and microphone and internet access to allow videoconferencing

Exclusion Criteria:

* They had consulted on the design and content of the intervention or study
* They have already participated in a substantial mindfulness-based course
* They are currently engaged or are planning to engage with another psychological intervention during the course of the study
* They currently engage in regular mindfulness-based practice
* They do not have the practical means and time available to be able to attend the intervention during the dates outlined on the information sheet and commit to at-home practice
* They have scores >19 on PHQ-8 (indicating 'severe' depressive symptom severity; Kroenke et al., 2009) or >15 on GAD (indicating 'severe' level of anxiety; Spitzer et al., 2006)
* They have a problem with alcohol or recreational drug misuse
* They have experienced thoughts about harming themselves or others in the last 12 months
* They have been given a diagnosis of psychosis
* They are currently experiencing high levels of distress and/or currently feeling particularly fragile
* They have experienced a bereavement of someone close to them in the last year or are continuing to experience continuing grief in relation to losing someone further back in time
* They have had traumatic experiences that they continue to be troubled by (including, but not limited to, receiving diagnosis of post-traumatic stress disorder)
* They experience significant difficulty being in a group with other people.

NB: for further details re the FAQL-PB and PHQ-8, please see the outcome measures section.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline at week 15 on the Food Allergy Quality of Life-Parental Burden scale - 17 item version (FAQL-PB) | Post intervention (week 15)
  This measures quality of life in parents of children with food allergies producing a score between 17 and 119, with higher scores indicating a greater burden on the family.

SECONDARY OUTCOMES:
Change from baseline at week 23 on the Food Allergy Quality of Life-Parental Burden scale - 17 item version (FAQL-PB) | Follow up (week 23)
  This measures quality of life in parents of children with food allergies producing a score between 17 and 119, with higher scores indicating a greater burden on the family.
Change from baseline at week 15 on the Generalized Anxiety Disorder screener - 7 items (GAD-7) | Post intervention (week 15)
  This measures symptoms of anxiety producing a score between 0 and 21, with higher scores indicating greater symptom severity.
Change from baseline at week 23 on the Generalized Anxiety Disorder screener - 7 items (GAD-7) | Follow up (week 23)
  This measures symptoms of anxiety producing a score between 0 and 21, with higher scores indicating greater symptom severity.
Change from baseline at week 15 on the Patient Health Questionnaire - 8 items (PHQ-8) | Post intervention (week 15)
  This measures symptoms of depression producing a score between 0 and 24, with higher scores indicating greater symptom severity.
Change from baseline at week 23 on the Patient Health Questionnaire - 8 items (PHQ-8) | Follow up (week 23)
  This measures symptoms of depression producing a score between 0 and 24, with higher scores indicating greater symptom severity.
Change from baseline at week 15 on the Perceived Stress Scale - 10 items (PSS) | Post intervention (week 15)
  This measures the perception of stress producing a score between 0 and 40, with higher scores indicating greater perceived stress.
Change from baseline at week 23 on the Perceived Stress Scale - 10 items (PSS) | Follow up (week 23)
  This measures the perception of stress producing a score between 0 and 40, with higher scores indicating greater perceived stress.
Change from baseline at week 15 on the Five-Facet Mindfulness Questionnaire - 15 items (FFMQ-15) | Post intervention (week 15)
  This measures trait mindfulness producing a score from 15 to 75, with higher score indicating greater trait mindfulness.
Change from baseline at week 23 on the Five-Facet Mindfulness Questionnaire - 15 items (FFMQ-15) | Follow up (week 23)
  This measures trait mindfulness producing a score from 15 to 75, with higher score indicating greater trait mindfulness.
Change from baseline at week 15 on the Perth Emotional Reactivity Scale Short Form - 18 items | Post intervention (week 15)
  This measures emotional reactivity producing separate composite scores for positive and negative emotion (i.e. 'general positive reactivity' and 'general negative reactivity'), each of which varies between 9 and 45, with higher scores indicating greater emotional reactivity. Note: this corrects a previous error where it was mistakenly stated that this scale produces a single overall score.
Change from baseline at week 23 on the Perth Emotional Reactivity Scale Short Form - 18 items | Post intervention (week 23)
  This measures emotional reactivity producing separate composite scores for positive and negative emotion (i.e. 'general positive reactivity' and 'general negative reactivity'), each of which varies between 9 and 45, with higher scores indicating greater emotional reactivity. Note: this corrects a previous error where it was mistakenly stated that this scale produces a single overall score.
Change from baseline at week 15 on the Leiden Index of Depression Sensitivity-Revised - 34 items | Post intervention (week 15)
  This measures cognitive reactivity producing a score between 0 and 136, with higher scores indicating greater cognitive reactivity.
Change from baseline at week 23 on the Leiden Index of Depression Sensitivity-Revised - 34 items | Post intervention (week 23)
  This measures cognitive reactivity producing a score between 0 and 136, with higher scores indicating greater cognitive reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Craig, MSc, Principal Investigator — Canterbury Christ Church University; Fergal Jones, PhD, PsychD, Study Director — Canterbury Christ Church University; Christina Jones, PhD, Study Director — University of Surrey
Locations (1):
- Salomons Institute for Applied Psychology, Royal Tunbridge Wells, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to other researchers on email request to the corresponding author after the study findings have been published in a peer reviewed journal.